CLINICAL TRIAL: NCT01298817
Title: Use of a Soy-based Meal Replacement Weight Loss Intervention to Impact Ectopic Fat and Associated Cardio-metabolic Risk in Obese, Older Adults: A Feasibility Study
Brief Title: Use of a Soy-based Meal Replacement Weight Loss Intervention to Impact Ectopic Fat
Acronym: SILVER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00015659
Record Dates: First submitted 2011-02-17; First posted 2011-02-18 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Abdominal Obesity
Keywords: Obesity; Aging; Soy; Weight Loss; Ectopic Fat
MeSH Terms: conditions — Obesity, Abdominal; Obesity; Weight Loss | interventions — Whey

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Soy, Prepared Meals (Experimental): Soy-based meal replacement weight loss group with additional meals provided
  Interventions: Dietary Supplement: Medifast meal replacement products
- Non soy prepared meals (Active Comparator): Non-soy based meal replacement weight loss group with additional meals provided
  Interventions: Dietary Supplement: Medifast meal replacement products

INTERVENTIONS:
Dietary Supplement: Medifast meal replacement products — A total of 4 meal replacement (MR)products per participant per day will be used. Approximately 2/3rd of the Medifast® MR product line is soy protein-based (i.e. at least 7 g of total protein coming from soy) with the remaining 1/3rd of items deriving total protein content from animal sources (whey and egg). The soy used in Medifast products is Solae SUPRO® water-washed soy protein isolate. Depending on seasonal variations, soy MR products contain approximately 1.5-3.0 milligrams of soy isoflavones for every 1 gram of soy protein. Thus, participants in the soy treatment arm will consume at least 28 g/soy protein and 42-108 mg/isoflavones per day.
  Other Names: Soy
  Arms: Soy, Prepared Meals
Dietary Supplement: Medifast meal replacement products — A total of 4 meal replacement (MR)products per participant per day will be used. Approximately 2/3rd of the Medifast® MR product line is soy protein-based (i.e. at least 7 g of total protein coming from soy) with the remaining 1/3rd of items deriving total protein content from animal sources (whey and egg). This group will receive the non soy supplements.
  Other Names: whey
  Arms: Non soy prepared meals

SUMMARY:
The main objectives of this study are to collect pilot data to assess feasibility (accrual, retention, compliance), to estimate the variability of outcome measures, and to obtain preliminary estimates of treatment efficacy based on group differences in body composition (decreases in ectopic fat stores while maintaining lean mass), cardio-metabolic risk factors including glucoregulatory function (glucose, insulin), inflammation (C-reactive protein, IL-6), blood pressure and lipids (HDL, LDL, TC, TG), and measures of physical function and muscle strength. While this is just a pilot study, randomization will be used so that the investigators can obtain a realistic estimate of accrual (which is often less in a randomized trial) and an unbiased estimate of treatment efficacy.

The investigators will accomplish these objectives by conducting a 2-arm, 3-month randomized, clinical trial in 24 older (60-79), abdominally obese (BMI ≥30 kg/m2 and waist circumference ≥ 102 cm and ≥ 88 cm in men and women, respectively) men and women. Participants will be randomized to a soy-based or animal-based, 3-month, hypocaloric dietary intervention to achieve our specific aims:

Primary Aim: To determine our ability to recruit and retain older, obese adults to a 3 month soy-based meal replacement weight loss intervention and assess the study participant's ability to adhere to the intervention protocol (weight, compliance logs, serum isoflavones).

Secondary Aims:

1. To estimate the variability of and obtain preliminary estimates of the effect of the soy-based meal replacement on measures of body composition, including abdominal (total, subcutaneous and visceral fat), liver, and pericardial fat; anthropometrics (body weight, waist/hip circumference); and whole body fat and lean mass.
2. To estimate the variability of and obtain preliminary estimates of the effect of the soy-based meal replacement on biomarkers of cardiometabolic risk including glucoregulatory function (glucose, insulin), inflammation (C-reactive protein, IL-6), blood pressure and lipids (HDL, LDL, TC, TG).
3. To estimate the variability of and obtain preliminary estimates of the effect of the soy-based meal replacement on physical function (short physical performance battery, 400-m walk) and muscle strength (grip and knee extensor strength) and size (CT thigh muscle).
4. To document any adverse events associated with the soy-based meal replacement.

ELIGIBILITY:
Inclusion Criteria:

* Age = 60-79 years old
* BMI ≥ 27 kg/m2
* Waist Circumference= men ≥ 102 cm; women ≥ 88 cm
* Non-impaired cognitive function (MMSE > 21)
* Willing to provide informed consent
* No contraindications for participation in weight loss
* Able to provide own transportation to study visits and intervention
* Willing to consume meal replacement products (i.e. no soy/dairy allergies, product found to be palatable)
* Not involved in any other research study

Exclusion Criteria:

* Weight loss or gain (±5%) in past 6 months
* Body mass > 136 kg (DXA limit)
* Regular smoker (> 1 cigarette/day) within past year
* History of alcohol or substance abuse or dependence within the past 2 years (DSM IV criteria)
* Insulin-dependent or uncontrolled diabetes (FPG ≥ 126 mg/dL)
* Self-reported hepatitis
* Abnormal kidney function (creatinine > 2.0)
* Abnormal liver blood test (AST, ALT, total bilirubin- greater than twice the upper limit of normal; albumin - less than 2.0)
* Unstable angina
* MI, PCI or cardiac surgery < 3 month ago
* Uncontrolled blood pressure (> 160/90 mmHg)
* Chronic pulmonary disease (> mild or recent exacerbations)
* Thyroid disease
* Known significant hematological disease (including HBG < 11)
* Active known cancer requiring treatment in past year (except non-melanoma skin cancers)
* Life expectancy < 2 years
* Regular use of any medications that could influence study variables (growth/steroid hormones, including estrogen replacements, thiazolidinediones, statins, regular anti-inflammatory medications, weight loss medications, etc.)

Ages: 60 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Protocol Compliance | Baseline, weekly (1 time per week for 11 weeks), and at 12 week follow-up
  To determine our ability to recruit and retain older, obese adults to a 3 month soy-based meal replacement weight loss intervention and assess the study participant's ability to adhere to the intervention protocol (weight, compliance logs, serum isoflavones).

SECONDARY OUTCOMES:
Change in Body Composition | Baseline and at the 12-week follow up
  To estimate the variability of and obtain preliminary estimates of the effect of the soy-based meal replacement on measures of body composition, including abdominal (total, subcutaneous and visceral fat), liver, and pericardial fat; anthropometrics (body weight, waist/hip circumference); and whole body fat and lean mass.
Change in Cardiometabolic Health | Baseline and at the 12-week follow up
  To estimate the variability of and obtain preliminary estimates of the effect of the soy-based meal replacement on biomarkers of cardiometabolic risk including glucoregulatory function (glucose, insulin), inflammation (C-reactive protein, IL-6), blood pressure and lipids (HDL, LDL, TC, TG).
Change in Physical Function | Baseline and at the 12 week follow up
  To estimate the variability of and obtain preliminary estimates of the effect of the soy-based meal replacement on physical function (short physical performance battery, 400-m walk) and muscle strength (grip and knee extensor strength) and size (CT thigh muscle).
Number of participants with adverse events as a measure of safety and tolerability | Baseline, weekly (1 time per week for 11 weeks), and at 12 week follow-up
  To document any adverse events associated with the soy-based meal replacement.

CONTACTS AND LOCATIONS:
Overall Officials: Mara Vitolins, DrPH, Principal Investigator — Wake Forest University
Locations (1):
- Wake Forest University, Winston-Salem, North Carolina, United States